CLINICAL TRIAL: NCT02658136
Title: Computed Tomography Estimated Right Ventricular Function and Exercise Capacity in Patients With Continuous-flow Left Ventricular Assist Devices
Brief Title: Right Ventricular Function and Exercise Capacity in Patients With Continuous-flow Left Ventricular Assist Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finn Gustafsson (Other)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, MD; PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 51347
Record Dates: First submitted 2016-01-12; First posted 2016-01-18 (Estimated); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 arm study: CCT estimated right ventricular function. (Other): By use of Cardiac computed tomography, the ejection faction of the right ventricle will be visualized and measured in all participants.
  Interventions: Other: Cardiac Computed tomography

INTERVENTIONS:
Other: Cardiac Computed tomography

SUMMARY:
Exercise capacity in continous-flow left ventricular assist device (CF-LVAD) patients remains severely reduced post-implant. While the effect of right ventricular (RV) failure early after pump implantation, and its effect on outcome has been extensively studied, the effects of late RV failure on exercise capacity and quality of life (QOL) has been sparsely described. Thus the purpose of this study is to examine RV function and the association to exercise capacity in CF-LVAD patients.

DETAILED DESCRIPTION:
When pharmacological therapy becomes insufficient in advanced end-stage heart failure (HF) transplantation remains the gold standard of therapies. However, due to a severe lack of donor organs, mechanical circulatory support is an alternative option for some eligible patients. Mechanical circulatory support in the form of a CF-LVAD is a pump supporting the left ventricle by pumping blood from the apex to the ascending aortae. Implantation with a CF-LVAD increases survival and improves quality of life, but peak oxygen uptake (peak VO2) remains severely reduced post-implant. Complex central and peripheral hallmarks of heart failure attribute to the continued work intolerance. Furthermore a fixed CF-LVAD pump speed prevents adequate circulatory support during strenuous exercise. The effects of late right ventricular (RV) failure on exercise capacity and quality of life (QOL) is, however, unknown and the purpose of this study is to examine RV function and the association to exercise capacity in CF-LVAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients from Department of Cardiology, Rigshospitalet, Denmark.
* Age ≥ 18 years.
* Ischemic or non-ischemic cardiomyopathy.
* Signed informed consent.

Exclusion Criteria:

* Unstable patients with the need for intravenous inotropic therapy.
* CF-LVAD implantation less than one month ago.
* eGFR < 45 ml/min.
* Contrast allergy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02; Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Rigshospitalet., Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Arm Study: CCT Estimated Right Ventricular Function.: Fifteen patients with HeartMate (HM) II or III underwent echocardiography and maximal cardiopulmonary exercise test. Subsequently, contrast-enhanced 4D Cardiac Computed Tomography(CCT) scans were performed at rest and immediately after two minutes of supine 25 Watt ergometer bike exercise.
Period: Overall Study
Arm/Group | 1 Arm Study: CCT Estimated Right Ventricular Function.
Started (Approved: 02-03-2016 (1-day study)) | 15 (Approved to start in year 2016. Goal was to reach 15 participants (1 day study).)
Completed | 15 (Date of end of study: June 2017, N=15)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 Arm Study: CCT Estimated Right Ventricular Function.: Cardiac Computed tomography
Arm/Group | 1 Arm Study: CCT Estimated Right Ventricular Function.
Number analyzed (Participants) | 15
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak Oxygen Uptake
Description: Cardiopulmonary exercise testing (CPET) measuring peak oxygen uptake in ml/kg/min.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Single-arm Study: Exercise and Right Ventricular Function in Patients With LVADs: Peak oxygen uptake (ml/kg/min) was measured on upright ergometer bicycle
Arm/Group | Single-arm Study: Exercise and Right Ventricular Function in Patients With LVADs
Number analyzed (Participants) | 15
ml/kg/min | 15 (5)

2. Secondary Outcome: Right Ventricular Function (RVEF) During Exercise
Description: Right ventricular function during exercise was estimated by use of contrast enhanced cardiac computed tomography.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: percent of ejected blood
Groups:
- CCT Estimated Right Ventricular Function.: Right ventricular ejection fraction was estimated by use of contrast-enhanced CCT in all study participants.
Arm/Group | CCT Estimated Right Ventricular Function.
Number analyzed (Participants) | 15
percent of ejected blood | 37 (8)

ADVERSE EVENTS:
Time Frame: Observed app. 1 hour after contrast infusion and > 30 min after each completed exercise test. No AE/SAE was observed.
Groups:
- 1 Arm Study: CCT Estimated Right Ventricular Function.: Fifteen patients with HeartMate (HM) II or 3 underwent echocardiography and maximal cardiopulmonary exercise test. Subsequently, contrast-enhanced four-dimensional (4D) cardiac computed tomography (CCT) scans were performed at rest and immediately after two minutes of supine 25 Watt ergometer bike exercise.
Arm/Group | 1 Arm Study: CCT Estimated Right Ventricular Function.
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT02658136/Prot_SAP_000.pdf